CLINICAL TRIAL: NCT03726970
Title: Effect of Metal Artifacts Reduction Protocols and Tube Potential Difference on Metal Artifacts in Cone Beam Computed
Brief Title: Effect of Metal Artifacts Reduction Orotocols and Electric Potential Difference on Metal Artifacts in Cone Beam Computed Tomography
Acronym: DTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marina Salib, Masters degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RAD
Record Dates: First submitted 2018-10-12; First posted 2018-11-01 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Metal Artifacts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tube Potential difference (Experimental): Different kVp values of the CBCT machine 70, 80 ,90 kVp
  Interventions: Radiation: CBCT radiation
- MAR tool (Experimental): MAR option in the software off and on
  Interventions: Radiation: CBCT radiation

INTERVENTIONS:
Radiation: CBCT radiation — CBCT scanning

SUMMARY:
The effect of metal artifacts reduction protocols and tube potential difference on the metallic artifacts in cone beam computed tomography

DETAILED DESCRIPTION:
Our study is a quantitative as well as a qualitative assessment of the metal artifacts in the CBCT images in a bio models with multiple adjacent dental implants and single isolated implants , while using different MAR protocols inherited in the CBCT soft ware , as well as change in the tube potential difference of the CBCT unit

ELIGIBILITY:
Inclusion Criteria:

* bio models of a lower jaw Titanium implants Porcelain fused to metal crowns

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Dental implant linear measurement | 1 month
  The implant length and width in millimeters will be assessed in the presence of the artifacts with and without the activation of the MAR tool of the CBCT soft ware, also change in the potential difference will be done with and without the activation of MAR tool

SECONDARY OUTCOMES:
Bone- implant interphase | 1 month
  Qualitative assessment if bone - implant interphase, will be either zero or 1 zero indicate that bone implant interphase cannot be assessed , one indicate that the bone implant interphase can be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mushira M Dahba, Doctorate, Study Director — Cairo University
Locations (1):
- Marina Salib, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided